CLINICAL TRIAL: NCT06502938
Title: To Evaluate Percutaneous Coronary Intervention Assisted by the Control System of Panvascular Interventional Surgery Efficacy and Safety Clinical Trials
Brief Title: A Clinical Trial Evaluating the Pan-vascular Interventional Robotic System for Panvascularization Interventional Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institute of Advanced Biomedical Robot Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ge Junbo, Chief of Cardiology, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPTAIN-C
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pan-vascular interventional robotic system group (Experimental): Pan-vascular interventional robotic system assisted PCI
  Interventions: Device: Pan-vascular interventional robotic system
- Artificial control group (Experimental): Traditional artificial percutaneous coronary intervention
  Interventions: Procedure: Traditional artificial percutaneous coronary intervention

INTERVENTIONS:
Device: Pan-vascular interventional robotic system — Pan-vascular interventional robotic system assited PCI for delivery and manipulation of guidewires, catheters, and quick exchange balloon dilatation catheters/stents.
  Arms: Pan-vascular interventional robotic system group
Procedure: Traditional artificial percutaneous coronary intervention — Doctors perform traditional percutaneous coronary intervention
  Arms: Artificial control group

SUMMARY:
The purpose of this prospective, randomized, open, parallel controlled, multicenter trial is to investigate the efficacy and safety of the pan-vascular interventional robotic system for percutaneous coronary intervention (PCI). Investigators will evaluate clinical success, technical success, and record intraoperative data (PCI time, total operating time, contrast agent dose, radiation exposure dose, etc.). All subjects were followed up on the day of surgery, before discharge and 1 month after surgery to observe the safety indicators.

ELIGIBILITY:
Inclusion Criteria:

1. General Inclusion criteria:

1. 18 years old ≤ age ≤85 years old;
2. have a clinical indication for PCI (clinical evidence of ischemic heart disease or a positive functional study);
3. Subject or guardian can understand the purpose of the experiment and sign informed consent voluntarily Book and willing to cooperate to complete the follow-up.

2. Angiographic inclusion criteria:

1. The stenosis degree of visual target lesion ≥50%;
2. 2.5mm≤ Visual target vessel diameter ≤4.0mm;
3. Visual target lesions ≤38mm in length, or successive small lesions that can be completely covered by a single stent;
4. Target lesions to be treated intraoperatively cannot be treated in stages.

Exclusion Criteria:

1. General exclusion criteria 1)A stroke occurred within 30 days prior to surgery; 2)Percutaneous coronary intervention was performed within 72 hours before surgery; 3)Acute myocardial infarction, cardiogenic shock, or infarction occurred within 48 hours before surgery Received CPR; 4)Other cardiac procedures (such as aortic valve placement) are scheduled within 30 days of surgery Coronary artery bypass grafting, etc.); 5)Pregnant or lactating female subjects; 6)Severe hepatic or renal insufficiency or bleeding tendency; 7)Known allergy to interventional device materials and their coatings, or allergy to contrast agents; 8)Severe stenosis, occlusion of blood vessels at the intended puncture site, or local skin infection and uncontrollable; 9)Are participating in other interventional clinical studies, and have not completed the evaluation of the primary endpoint of the relevant study; 10)Participants who had other contraindications for interventional therapy or were judged by the investigator to be unsuitable for participation in the study;
2. Angiographic exclusion criteria 1)The TIMI blood flow grade of the target lesion was < 2; 2)Treatment requiring intrastent restenosis, or prior placement of a stent in the target vessel near both ends of the target lesion; 3)Severe tortuosity or severe calcification of blood vessels; 4)There's an intracavitary thrombus; 5)In addition to balloon forming and stent implantation, other treatments (such as atheromatectomy, rotary grinding, laser ablation, etc.) are also required at the same time; 6)The researchers determined that percutaneous coronary intervention was not suitable for robotic assistance or that there might be high risks in the process.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | Immediate postoperative angiography
  Immediate postoperative angiography showed residual stenosis < 30% and TIMI blood flow fraction Level 3.
Clinical Success | Discharge or 48 hours post intervention, whichever comes first
  No MACE occurred in hospital.

SECONDARY OUTCOMES:
Technical success rate | Procedure
  1. PCI was assisted by the Pan-vascular Interventional Robotic System.
  2. No unplanned complete conversion to artificial surgery occurred due to the inability to complete the delivery of the guide wire or balloon/stent catheter through the vessel with the test instrument as intended, or due to insufficient guide catheter support.
Radiation Exposure | Procedure
  Patient and Main operator radiation exposure dose recorded by portable radiation
Fluoroscopy Time | Procedure
  Total Fluoroscopy Time during procedure will be captured.
Contrast agent dosage | Procedure
  The total amount of contrast agent used during the whole procedure.
Procedure Time | Procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
PCI time | Procedure
  Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
the Pan-vascular Interventional Robotic Systemt performance evaluation | After the operation
  The performance of the product was subjectively evaluated by the surgeon.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital,Sun Yat-sen University, Guanzhou, Guandong
  - Linfen Central Hospital, Shanxi, Linfen
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang